CLINICAL TRIAL: NCT02893709
Title: Factors Influencing the Human Gut Microbiome Profile in Multi-ethnic Groups of the Singapore Community (FAMES)
Acronym: FAMES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changi General Hospital (Other)
Collaborators: National University of Singapore (Other); Universiti Teknologi Mara (Other)
Responsible Party: Principal Investigator, Ang Tiing Leong, Senior Consultant Gastroenterologist, Changi General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FAMES
Record Dates: First submitted 2016-08-24; First posted 2016-09-08 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Omeprazole (Experimental): A course of omeprazole at therapeutic dose (20 mg daily) for a duration of 7 days
  Interventions: Drug: Omeprazole

INTERVENTIONS:
Drug: Omeprazole — Oral administration of omeprazole at therapeutic dose (20 mg daily) for a duration of 7 days
  Other Names: Omezole20

SUMMARY:
The objectives of this study are to examine the effects of ethnicity, gender, and proton pump inhibitor (PPI, omeprazole), on the human gut microbiome. The investigators hypothesize that PPI therapy might perturb microbial communities and alter the gut microbiome. Young, healthy subjects of Chinese, Malay and Indian ancestry, were enrolled. They were required to provide a baseline stool sample (Day 1) and were then given a course of omeprazole at therapeutic dose (20 mg daily) for a duration of 7 days. Stool samples were collected again on Day 7 and Day 14 (one week after stopping omeprazole). The DNA samples were subjected to 16S ribosomal ribonucleic acid (rRNA) sequencing.

DETAILED DESCRIPTION:
Background and Aim: The objectives of this study are to examine the effects of ethnicity, gender, and proton pump inhibitor (PPI, omeprazole), on the human gut microbiome. PPIs are commonly used for the treatment of acid-related disorders. The investigators hypothesize that PPI therapy might perturb microbial communities and alter the gut microbiome.

Methods: Healthy subjects of Chinese (n=12), Malay (n=12) and Indian (n=10) ancestry, aged 21-37 years old, were enrolled. They were required to provide a baseline stool sample (Day 1) and were then given a course of omeprazole at therapeutic dose (20 mg daily) for a duration of 7 days. Stool samples were collected again on Day 7 and Day 14 (one week after stopping omeprazole). Microbial DNA was extracted from the stool samples. This was followed by PCR, library construction, 16S rRNA sequencing using Illumina MiSEQ, and statistical and bioinformatics analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed written informed consent,
2. Aged between 21-35 years of age,
3. Chinese, Malay or Indian ancestry through three generations,
4. Clinical laboratory assessment results within normal limits, unless the deviation is considered not clinically significant by the investigator,
5. Subject is healthy with no clinically significant disease or condition as determined through their medical history, physical examination, and results from clinical laboratory tests that are performed within 2 weeks before the baseline visit at Day 1,
6. Ability to communicate with the investigator and to understand and comply with all requirements of study participation.
7. Female subjects must be in the first half of their menstrual cycle (i.e. 1 to 14 days after the end of the previous menstruation) at Research Study entry.

Exclusion Criteria:

1. Any acute illness within 2 weeks before Day 1, unless otherwise approved by the PI,
2. Presence of chronic illnesses e.g. diabetes, renal disease, gastrointestinal disease, etc., which, in the opinion of the investigator, could compromise the data of the study,
3. Subjects who declare themselves positive for HIV or viral hepatitis (Hepatitis A, B, C),
4. Treatment within the previous 3 months with antibiotics,
5. Treatment with any prescription or over-the-counter (OTC) medications, or herbal supplements within 4 weeks of Day 1 unless approved by the PI,
6. Consumption of probiotics or lactobacillus-containing products e.g. Yakult, Vitagen or Yogurt within 4 weeks of Day 1 unless approved by the PI,
7. Abnormal biochemistry indicators,
8. Poor peripheral venous access,
9. Involvement in the planning or conduct of this study,
10. Irregular bowel habits or complains of constipation problem.

Ages: 21 Years to 37 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2015-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change in species diversity after omeprazole treatment, as measured by diversity indices | 1 week, 2 weeks
Emergence of signature taxa after omeprazole treatment, as measured by indicator value | 1 week, 2 weeks
Differences in species diversity between gender, as measured by diversity indices | Baseline
Differences signature taxa among ethnic groups, as measured by indicator value | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Tiing Leong Ang, MD, Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Freedberg DE, Toussaint NC, Chen SP, Ratner AJ, Whittier S, Wang TC, Wang HH, Abrams JA. Proton Pump Inhibitors Alter Specific Taxa in the Human Gastrointestinal Microbiome: A Crossover Trial. Gastroenterology. 2015 Oct;149(4):883-5.e9. doi: 10.1053/j.gastro.2015.06.043. Epub 2015 Jul 9. PMID 26164495
- [Background] Jackson MA, Goodrich JK, Maxan ME, Freedberg DE, Abrams JA, Poole AC, Sutter JL, Welter D, Ley RE, Bell JT, Spector TD, Steves CJ. Proton pump inhibitors alter the composition of the gut microbiota. Gut. 2016 May;65(5):749-56. doi: 10.1136/gutjnl-2015-310861. Epub 2015 Dec 30. PMID 26719299
- [Background] Clooney AG, Bernstein CN, Leslie WD, Vagianos K, Sargent M, Laserna-Mendieta EJ, Claesson MJ, Targownik LE. A comparison of the gut microbiome between long-term users and non-users of proton pump inhibitors. Aliment Pharmacol Ther. 2016 May;43(9):974-84. doi: 10.1111/apt.13568. Epub 2016 Feb 29. PMID 26923470
- [Background] Imhann F, Bonder MJ, Vich Vila A, Fu J, Mujagic Z, Vork L, Tigchelaar EF, Jankipersadsing SA, Cenit MC, Harmsen HJ, Dijkstra G, Franke L, Xavier RJ, Jonkers D, Wijmenga C, Weersma RK, Zhernakova A. Proton pump inhibitors affect the gut microbiome. Gut. 2016 May;65(5):740-8. doi: 10.1136/gutjnl-2015-310376. Epub 2015 Dec 9. PMID 26657899